CLINICAL TRIAL: NCT05033613
Title: Home Blood Pressure Monitoring Before and After COVID-19 Vaccination in Patients at High Risk of Cardiovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202107076RINA
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Pain; Fatigue; Headache; Myalgia; Chills; Arthralgia; Fever
Keywords: COVID-19 vaccination, Side effects
MeSH Terms: conditions — Pain; Fatigue; Headache; Myalgia; Chills; Arthralgia; Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: heart rate、arrhythmia、blood pressure、central body temperature (ear temperature) and blood oxygen saturation level. — heart rate、arrhythmia、blood pressure、central body temperature (ear temperature) and blood oxygen saturation level.

SUMMARY:
The coronavirus SARS-CoV-2 causing COVID-19 was pandemic since 2020. Vaccination is one of the most important measure to control the outbreak. The countries of the world started the vaccination since December, 2020. Taiwan started since March, 21st, 2021. Currently, Taiwanese people receive COVID-19 vaccination by either AZ or Moderna; Pfizer/BNT vaccine may import in the near future. The side effects post vaccination including injection site pain, fatigue, headache, myalgia, chills, arthralgia, fever, and so on. Incidence of side effects more frequent in young people than elders; more frequent in the first dose than second dose in AZ vaccine; more frequent in the second dose in Moderna or Pfizer/BNT vaccine. Taiwan V-watch is a system monitored by CDC for people proactive notification of side effects post COVID-19 vaccination. But it doesn't include the objective cardiovascular parameters, for example, heart rate, arrhythmia, blood pressure, central body temperature (ear temperature) and blood oxygen saturation level.

This study aims to monitor the physiologic and psychologic effects, and side effects before and after COVID-19 vaccination in patients at high cardiovascular risk, including hypertension, hyperlipidemia, and type 2 diabetes, and arrhythmia or coronary artery disease. The investigators arrange two weeks of continuous home BP/HR monitoring (7 days pre- and post-vaccination) for evaluation of physiologic effects post vaccination. Due to fever noted in some people post-vaccination, the investigators also measure ear temperature, pulse oximetry, and environmental temperature and humidity, for the reference of BP monitoring.

In conclusion, this study may provide important information of cardiovascular response and psychosocial effects after SARS-CoV-2 vaccination for proactive prevention of cardiovascular complications.

ELIGIBILITY:
Inclusion Criteria:

* People at high cardiovascular risk.
* Clinical diagnosis of hypertension
* Clinical diagnosis of hyperlipidemia
* Clinical diagnosis of type 2 diabetes
* Clinical diagnosis of arrhythmia
* Clinical diagnosis of coronary artery disease
* Patients at the cardiology clinic.

Exclusion Criteria:

* People who have been diagnosed by a doctor as unsuitable for vaccination.
* People with serious injuries or catastrophic illness, such as cancer patients.
* People who stay in bed for a long time and cannot take care of themselves.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients at high cardiovascular risk, including hypertension, hyperlipidemia, and type 2 diabetes, and arrhythmia or coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-12-29 (Estimated); Study Completion 2022-12-29 (Estimated)

PRIMARY OUTCOMES:
Compare the physiological effects of different type of COVID-19 vaccines | From 1 Sep. 2021 to 1 Dec. 2022
  Compare the physiological effects of different type of COVID-19 vaccines, including cardiovascular aspects, blood pressure, heartbeat, blood oxygen, whether there is arrhythmia, whether there are changes in blood oxygen concentration and core body temperature (ear temperature).
Compare whether the subjective side effects of different type of COVID-19 vaccines are different | From 1 Sep. 2021 to 1 Dec. 2022
  Compare whether the subjective side effects of different type of COVID-19 vaccines are different, including fever, headache, dizziness, drowsiness, insomnia, palpitations, arrhythmia, nausea, vomiting, tiredness, pain, redness, heat or swelling at the injection site, difficulty breathing, muscles soreness, muscle weakness, abdominal pain, diarrhea, etc.
Compare the psychological stress effects of different type of COVID-19 vaccines | From 1 Sep. 2021 to 1 Dec. 2022
  Compare the psychological stress effects of different type of COVID-19 vaccines, choose to use the CES-D (The Center for Epidemiologic Studies Depression Scale) Questionnaire and PSQI (The Pittsburgh Sleep Quality Index), to measure and check whether there are differences.

CONTACTS AND LOCATIONS:
Overall Officials: TA-CHEN SU, Doctor, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Chung-Shan, Taiwan